CLINICAL TRIAL: NCT00286598
Title: Feet First: Increasing Activity Without Increasing the Risk of Foot Ulcers in People With Diabetes and Insensate Feet
Brief Title: Feet First: Promoting Physical Activity Among People With Diabetes Mellitus and Insensate Feet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UMHS IRB 1040047
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus; Peripheral Neuropathies
Keywords: foot ulcer; diabetes mellitus; motor activity; randomized controlled trial; prevention
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases; Foot Ulcer; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Feet First (Experimental): Phase 1: (enrollment to 3 months) 8 sessions with a physical therapist learning leg strengthening and balance exercises, and initiating a walking program Phase 2: Motivational enhancement calls from a nurse every 2 weeks.
  Interventions: Behavioral: Feet First
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Feet First — Phase 1: (enrollment to 3 months) 8 sessions with a physical therapist learning leg strengthening and balance exercises, and initiating a walking program Phase 2: Motivational enhancement calls from a nurse every 2 weeks.
  Arms: Feet First

SUMMARY:
The role of weight-bearing physical activity in the development of diabetic foot ulcers remains poorly understood. Regular participation in moderately intense physical activity (e.g. brisk walking ) reduces 8-year cardiovascular mortality in those with diabetes mellitus by over 30%. The American Diabetes Association (ADA) recommends at least 30 minutes of daily moderate intensity activity for people with diabetes. However, the ADA recommends that people with diabetes and insensate feet, which affects up to 40% of those with diabetes, should limit their walking because of concerns that walking could increase the risk of foot ulcers and amputation. Firm evidence is lacking to support these concerns; in fact, while a research fellow I conducted an observational study that showed daily weight-bearing activity may reduce the risk of foot ulceration among people with diabetic foot problems. A controlled clinical trial is needed to study these issues further.

The present study is a randomized controlled trial in 100 older adults with diabetes and insensate feet, 50 of whom will participate in an individually-tailored behavior-change intervention called "Feet First", and 50 of whom will be controls. The intervention is based on the extensively-tested CHAMPS model used by the Robert Wood Johnson Foundation's Active for Life Program. Feet First extends the target population beyond older adults generally to people with insensate feet due to diabetic peripheral neuropathy.

The specific aims of the study are:

* To determine whether Feet First intervention subjects achieve a greater increase in weight-bearing activity than control subjects, and
* To obtain preliminary evidence on intervention subjects' foot outcomes (foot function, foot-related self-care, and risk of foot ulcers), compared to control subjects.

DETAILED DESCRIPTION:
Physical activity is a vital component of self-management for patients with diabetes mellitus, yet there are special problems in patients whose disease is complicated by insensate feet (i.e. loss of protective sensation caused by diabetic distal symmetric sensory peripheral neuropathy). Foot ulcers develop in 15% of the 17 million people in the United States with diabetes mellitus, and contribute to 84% of foot or toe amputations. Foot ulcer risk is very high among those with insensate feet. Although the roles of neuropathy, plantar foot pressure, and footwear in foot ulcers have been extensively studied, the independent role of physical activity has not. The overall goal of this study is to determine whether a "lifestyle" physical activity intervention, based on the Second Community Healthy Activities Model Program for Seniors (CHAMPS II), which we call FEET FIRST, can be used to safely increase moderate-intensity physical activity (achieving at least 40% of maximal oxygen consumption, as in walking briskly) among people with diabetes and insensate feet. "Lifestyle" physical activity interventions help participants to accumulate at least 30 minutes of self-selected activities in short bouts during the day. CHAMPS II effectively and safely increased physical activity in sedentary older adults with multiple chronic illnesses.

Substantial research has also found that people with diabetic peripheral neuropathy are also at increased risk of falls. Diabetic peripheral neuropathy also leads to postural instability, i.e. impairment in measures of functional dynamic balance. Moreover, this instability worsens with age. People with diabetic peripheral neuropathy in particular tend to have ankle instability due to decreased proprioception, making them less able to rapidly recover balance during sudden ankle dorsiflexion, inversion or eversion when walking on uneven surfaces.

There is ample evidence that promotion of an active lifestyle and specific exercises targeting endurance, strength and balance improves reduces functional decline in the elderly, and that home-based exercise programs effectively decrease fall risk in the elderly as well. One small, non-randomized trial found preliminary evidence that a 3-week intervention that focused on ankle strength improved balance measures in those with diabetic peripheral neuropathy. However, no randomized studies have investigated the effect of a physical activity intervention on fall risk in community-dwelling people with diabetic peripheral neuropathy, who may also be at increased risk of cutaneous injuries (i.e. foot lesions) during weight-bearing activity. Before we unequivocally recommend to people with diabetic peripheral neuropathy that they engage in exercise, we need to determine that this will be safe for their feet, and not increase fall risk.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 1 or 2 diabetes mellitus
* Age 50 years or older
* Absent 5.07 Semmes Weinstein monofilament sensation to > 1 point on both feet
* Residence within 50 miles of Columbia, MO
* Functioning telephone service
* Not currently participating in 20 or more minutes of moderately intense activity more than twice a week

Exclusion Criteria:

* Hospitalization in the last year for any of the following reasons:
* Proliferative diabetic retinopathy
* Accelerated hypertension (systolic BP >200 or diastolic BP > 120)
* Myocardial infarction or unstable angina
* New hemodynamically significant arrhythmia
* Acute congestive heart failure
* Failure to attend 3 of the last 5 scheduled clinic visits
* Foot deformities requiring a custom shoe
* "Timed Up and Go" test 3 > 15 seconds Subjects unable to ambulate without assistance
* Severe cardiac autonomic neuropathy
* Lower extremity amputation > one digit
* Heart, kidney or other transplant
* Currently unhealed foot ulcer (or healed for less than 1 month

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2005-01; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change in weight-bearing physical activity (steps/day) | Baseline, 3, 6 and 12 months post-enrollment

SECONDARY OUTCOMES:
Partial or greater depth foot ulcer (Wagner Gr. 1 or deeper) | continuously post-enrollment for 12 months
Falls | continuously post-enrollment for 12 months
Self-reported foot disability | baseline, 6 and 12 months post enrollment
Foot-related self-care | baseline, 6 and 12 months post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W LeMaster, MD, MPH, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kruse RL, Lemaster JW, Madsen RW. Fall and balance outcomes after an intervention to promote leg strength, balance, and walking in people with diabetic peripheral neuropathy: "feet first" randomized controlled trial. Phys Ther. 2010 Nov;90(11):1568-79. doi: 10.2522/ptj.20090362. Epub 2010 Aug 26. PMID 20798179